CLINICAL TRIAL: NCT00016393
Title: A Phase II Trial of Epothilone B Analogue BMS-247550 (NSC #710428) (IND 59699) Administered Every 21 Days in Patients With Hormone Refractory Prostate Cancer
Brief Title: BMS-247550 in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068629; SWOG-S0111
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of BMS-247550 in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the prostate-specific antigen response to BMS-247550 in patients with hormone-refractory prostate cancer.
* Determine the overall survival and progression-free survival rate in patients treated with this drug.
* Determine the objective response rate (confirmed and unconfirmed complete and partial responses) in those patients with measurable disease treated with this drug.
* Evaluate the qualitative and quantitative toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive BMS-247550 IV over 3 hours on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses beyond CR.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 25-45 patients will be accrued for this study within 5-9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Stage D1 or D2 disease (T4, N0, M0; any T, N1-3, M0; or any T, any N, M1)
* Unresponsive or refractory to prior hormonal therapy by at least 1 of the following:

  * Progression of unidimensionally measurable lesion outside of a prior radiation port
  * Progression of non-measurable disease (e.g., bone scan)
* Rising prostate-specific antigen (PSA) on at least 2 consecutive measurements taken at least 7 days apart
* PSA at least 5 ng/mL
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL OR
* Creatinine clearance at least 40 mL/min

Other:

* No other malignancy within the past 5 years except adequately treated squamous cell or basal cell skin cancer, any carcinoma in situ, or stage I or II cancer in complete remission
* No other concurrent significant active illness that would preclude study participation
* Recovered from major infections
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 28 days since prior biologic therapy and recovered
* No more than 1 prior biologic (non-cytotoxic) therapy
* No concurrent biological response modifiers

Chemotherapy:

* No prior chemotherapy for this disease
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics
* At least 28 days since prior flutamide or ketoconazole
* At least 42 days since prior bicalutamide or nilutamide
* No concurrent hormonal therapy, except luteinizing hormone-releasing hormone therapy
* No concurrent corticosteroids

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy to less than 30% of bone marrow allowed
* No prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* At least 28 days since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery:

* Recovered from prior surgery
* Prior orchiectomy allowed

Other:

* No concurrent unconventional therapy (e.g., St. John's Wort, PC-SPES, or other herbal remedy for prostate cancer)
* Not planning to begin bisphosphonate therapy (patients already receiving bisphosphonates are eligible provided they have progressive disease)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hadi A. Hussain, MD, Study Chair — University of Michigan Rogel Cancer Center; Primo N. Lara, MD — University of California, Davis
Locations (28):
- United States (28):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Danville Radiation Therapy Center, Memphis, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Veterans Affairs Medical Center - Amarillo, Amarillo, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Hussain M, Tangen CM, Lara PN Jr, Vaishampayan UN, Petrylak DP, Colevas AD, Sakr WA, Crawford ED; Southwest Oncology Group. Ixabepilone (epothilone B analogue BMS-247550) is active in chemotherapy-naive patients with hormone-refractory prostate cancer: a Southwest Oncology Group trial S0111. J Clin Oncol. 2005 Dec 1;23(34):8724-9. doi: 10.1200/JCO.2005.02.4448. PMID 16314632